CLINICAL TRIAL: NCT06254027
Title: Multicentric, Randomized, Evaluator Blinded Clinical Investigation for the Evaluation of Efficacy and Safety of Two Medical Devices for the Treatment of Onychomycosis
Brief Title: Clinical Investigation for the Evaluation of Efficacy and Safety of Two Medical Devices for Onychomycosis Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Oystershell NV (Industry)
Collaborators: Eurofins (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23E3473
Record Dates: First submitted 2024-01-16; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-01

CONDITIONS: Onychomycosis
MeSH Terms: conditions — Onychomycosis | interventions — amorolfine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinded evaluation is done by digital analysis of photographs of the infected toenail or fingernail.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Forte (Experimental): Device:
  One application per day for 9 months.
  Interventions: Device: Forte
- Active Cover Light (Experimental): Device:
  One application per day for 9 months.
  Interventions: Device: Active Cover Light
- Loceryl 5% (Active Comparator): Drug: Loceryl 5% One application per week for 3 months
  Interventions: Drug: Loceryl

INTERVENTIONS:
Device: Forte — One application per day for a complete treatment period.
  Other Names: Excilor
  Arms: Forte
Device: Active Cover Light — One application per day for a complete treatment period.
  Other Names: Nailner
  Arms: Active Cover Light
Drug: Loceryl — One application per week for a complete treatment period.
  Other Names: Amorolfine
  Arms: Loceryl 5%

SUMMARY:
The goal of this clinical trial is to evaluate the effectiveness of FORTE, ACTIVE COVER LIGHT and Loceryl® in the treatment of onychomycosis based on the blinded evaluation of the percentage of healthy nail surface compared to baseline.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the effectiveness of FORTE (X92001873), ACTIVE COVER LIGHT (X92001872) and Loceryl® in the treatment of onychomycosis based on the blinded evaluation of the percentage of healthy nail surface compared to baseline.

The secondary objectives are to evaluate:

* Their effectiveness in the treatment of onychomycosis based on the microbiological cure (KOH staining and fungal culture)
* Their effectiveness in the improvement of nail appearance (onychomycosis evolution, onycholysis, dystrophy, discoloration, and nail thickening)
* Their effectiveness in the improvement of the quality of life of the patients using a specific questionnaire.
* Their effectiveness, tolerance and acceptability based on patient's opinion.
* Their safety The aim of the study is to demonstrate non-inferiority of the change in healthy nail surface from baseline to D270 of each product (μD) versus a predefined limit of 16% (clinically meaningful: μC) with a non-inferiority margin of δ = -5%

ELIGIBILITY:
Inclusion Criteria:

1. Patient having given freely her/his informed, written consent.
2. Patient having a good general health.
3. Age: more than 18 years.
4. Patient with superficial onychomycosis on at least one great toenail or fingernail (for at least 10% in each arm) or light to moderate disto-lateral onychomycosis (without matrix involvement and involvement <2/3 of the tablets).
5. Patient with positive KOH staining.
6. Patient cooperative and aware of the products modalities of use and the necessity and duration of the controls so that perfect adhesion to the protocol can be expected.
7. Patient being psychologically able to understand information and to give their/his/her consent.
8. Patient having stopped any systemic antifungal treatment since at least 6 months before screening.
9. Patient having stopped any topical antifungal treatment since at least 3 months before screening.
10. Patient who agrees to refrain from receiving pedicure/manicure, artificial nails and/or cosmetic nail varnish or other medication on the nail being treated for the entire study duration.
11. Female of childbearing potential should use a contraceptive regimen recognized as effective since at least 12 weeks before screening visit, during all the study and at least 1 month after study end.

Exclusion Criteria:

1. Pregnant, breastfeeding woman or woman planning a pregnancy during the study.
2. Patient considered by the investigator likely to be non-compliant with the protocol.
3. Patient enrolled in another clinical trial or which exclusion period is not over.
4. Patient with a condition or receiving a medication which, in the investigator's judgment, put the patient at undue risk.
5. Patient suffering from a severe or progressive disease (to investigator's discretion) such as uncontrolled diabetes, peripheral circulatory disease, HIV, psoriasis, lichen planus, immunosuppressive pathology…
6. Patient having a known allergy or hypersensitivity to one of the constituents of the tested products.
7. Patient with cutaneous pathology on studied zone (other than onychomycosis like angioma, dermatitis…).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of healthy surface (Performance) | 270 days
  Variation of the percentage of healthy surface after 270 days (9 months) of treatment with the test medical devices (FORTE or ACTIVE COVER LIGHT) or reference product (Loceryl) versus baseline value.

SECONDARY OUTCOMES:
Percentage of healthy surface (Performance) | 30 days; 90 days; 180 days
  Variation of the percentage of healthy nail surface versus baseline value.
Microbiological efficacy: KOH staining (Performance) | 270 days (month 9)
  Evaluation of microbiological efficacy versus baseline by KOH staining and fungal culture.
Clinical efficacy: Visual appearance of nail (including onycholysis, nail dystrophy, nail discoloration and nail thickening) (Performance) | Baseline, 30 days; 90 days, 180 days; 270 days
  Evaluation of the visual appearance of the nail by assessing following parameters: onycholysis, nail dystrophy, nail discoloration, and nail thickening by the investigator in live.
  Each parameter is scored from 0 (none) - 4 (severe). The total score of all parameters is an indication of the visual appearance of the nail.
Clinical efficacy: onychomycosis evolution (Performance) | 30 days; 90 days; 180 days; 270 days
  Assessment of onychomycosis evolution by the investigator in live by scoring:
  1. - Failure: increase in the total infected area or aggravation
  2. - Status Quo
  3. - Improvement: decrease of the total infected area
  4. - Success: Disappearance of the total infected area
Impact on quality of life (Performance) | Baseline, 30 days; 90 days, 180 days; 270 days
  Evaluation of the impact on the quality of life (QoL) of patients using a validated questionnaire (NailQoL).
  The questionnaire contains 15 questions, each using the scoring:
  * 0 (never)
  * 25 (rarely)
  * 50 (sometimes)
  * 75 (often)
  * 100 (all the time)
Subjective evaluation questionnaire for the patient (Performance) | 14 days; 30 days; 90 days; 180 days; 270 days
  Evaluation of efficacy, tolerance, and acceptability of the test medical devices and reference by the patients using a subjective evaluation questionnaire.
  The subjective evaluation questionnaire uses a scoring (Completely Agree, Agree, Neutral, Disagree or Completely disagree) or uses 'Yes/No'- questions to be able to provide a score for performance.
  Some open questions are added to allow the patients to elaborate on certain answers in order to have a better understanding of their response.
Evaluation of tolerance | 30 days; 90 days; 180 days; 270 days
  Evaluation of tolerance of the test medical devices and reference. Assessment is performed by the investigator via clinical evaluation and subject interrogation. The investigator will assign a score between 0 (bad tolerance) to 3 (very good tolerance).